CLINICAL TRIAL: NCT01785784
Title: Phase IV Clinical Trial of rhGM-CSF Hydro-gel for Topical Application on Deep 2nd Partial Thickness Burn
Brief Title: Efficacy and Safety Study of rhGM-CSF Gel to Treat Deep 2nd Thickness Burn
Acronym: rhGM-CSF
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Changchun GeneScience Pharmaceutical Co., Ltd. (Industry)
Collaborators: Shanghai Jiao Tong University School of Medicine (Other); Beijing Children's Hospital (Other); Third Military Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GenSci-002-CT
Record Dates: First submitted 2013-01-28; First posted 2013-02-07 (Estimated); Last update posted 2013-02-07 (Estimated); Status verified 2013-02

CONDITIONS: Deep Partial Thickness Burn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- burn patients (Experimental)
  Interventions: Drug: rhGM-CSF Gel

INTERVENTIONS:
Drug: rhGM-CSF Gel

SUMMARY:
This was a multicenter, randomized, phase Ⅳ study, to investigate the extensive efficacy and safety of Recombinant Human Granulocyte/Macrophage Colony-stimulating Factor Hydro-gel for Topical Application (rhGM-CSF Gel) on deep 2nd burn.

There are two parts of the phase Ⅳstudy, the first part was a multicenter, randomized, reference controlled study, all the subjects were randomized into two groups, test group (rhGM-CSF Gel) and control group (iodophor gauze), totally 358 deep 2nd burned patients were enrolled in first part of the study, 177 cases were enrolled in test group and 181 cases were enrolled in reference control group. In the test group, after the patients were enrolled in the group, clean the wound surface regularly and wash with normal saline, spread the test drug on the wound surface, bandaging with sterilized vaseline gauze, change the drug product every two or one day according to the effusion. In the reference control group, after the patients were enrolled in the group, clean the wound surface regularly and wash with normal saline, bandaging with iodophor gauze, change the drug product every two or one day according to the effusion. Whole treatment were lasted till the wound surface was healing completely, if it is not recovered in 4 weeks, calculate and record the healing rate. The secondary part of the study was a multicenter, open study, to investigate the safety of rhGM-CSF on deep 2nd burn patients. Totally 2329 patients were enrolled in this part of the study.

ELIGIBILITY:
Inclusion Criteria:

* age is not less than 3 years old, any gender is ok.
* the subject who is diagnosed as deep 2nd thickness burn
* the subject who was not administrated with any other topical durg on wound surface before enrolled in the clinical study.
* the subject who sign the <informed consent>

Exclusion Criteria:

* age is less than 3 years old
* the subject who participated in any other clinical trial within 3 months
* the subject who was administrated with any other topical drug on wound surface before enrolled in the clinical study
* the female subject who is in lactation or pregnancy
* the subject who are allergic to rhGM-CSF, or has the allergic history to many drug products or has the allergic disease recently
* the subject who has serious heart disease, unstable angina pectoris break out, cardiac functional insufficiency, myocardial infarction or serious general infection.
* the subject who has serious renal inadequacy, creatinine(Cr) is more than 2.5 times of the upper limit
* aspartate aminotransferase or alanine transpeptidase is more than 2.5 times of the upper limit
* the subject who use immunosuppressant

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2510 (Actual)
Dates: Start 2010-11; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

PRIMARY OUTCOMES:
100% healing time of the wound surface | 4 weeks

SECONDARY OUTCOMES:
appearance of the wound surface | day 0, day 2, day 4, day 6, day 8, day 10, day 12, day 14, day16, day 18, day 20, day 22, day 24, day 26, day 28
  If the 100% healing date of the wound surface is less than 28 days, record the result until the 100% healing day.
healing rate of the wound surface | Day 8, day 10, day 12, day14, day 16, day 18, day 20, day22, day 24, day26 and day 28
  If the 100% healing date of the wound surface is less than 28 days, record the result until the 100% healing day.

OTHER OUTCOMES:
Heart Rate | day 0, day 2, day 4, day 6, day 8, day 10, day 12, day 14, day16, day 18, day 20, day 22, day 24, day 26, day 28
  If the 100% healing date of the wound surface is less than 28 days, record the result until the 100% healing day.
Body Temperature | day 0, day 2, day 4, day 6, day 8, day 10, day 12, day 14, day16, day 18, day 20, day 22, day 24, day 26, day 28
  If the 100% healing date of the wound surface is less than 28 days, record the result until the 100% healing day.
Blood Pressure | day 0, day 2, day 4, day 6, day 8, day 10, day 12, day 14, day16, day 18, day 20, day 22, day 24, day 26, day 28
  If the 100% healing date of the wound surface is less than 28 days, record the result until the 100% healing day.
Breathing Rate | day 0, day 2, day 4, day 6, day 8, day 10, day 12, day 14, day16, day 18, day 20, day 22, day 24, day 26, day 28
  If the 100% healing date of the wound surface is less than 28 days, record the result until the 100% healing day.
Blood Routine | day 0, day 28
  Blood routine should be tested before administration and after the last administration. If the 100% healing date of the wound surface is less than 28 days, record the result in the 100% healing day.
Urine Routine | day 0, day 28
  Urine routine should be tested before administration and after the last administration. If the 100% healing date of the wound surface is less than 28 days, record the result in the 100% healing day.
liver Function | day 0, day 28
  Liver function should be tested before administration and after the last administration. If the 100% healing date of the wound surface is less than 28 days, record the result in the 100% healing day.
Renal Function | day 0, day 28
  Renal function should be tested before administration and after the last administration. If the 100% healing date of the wound surface is less than 28 days, record the result in the 100% healing day.

CONTACTS AND LOCATIONS:
Overall Officials: Liao Zh Jiang, Doctor, Principal Investigator — Affiliated Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine